CLINICAL TRIAL: NCT03807323
Title: New Tools for Lasting Lifestyle Changes Among Inactive Obese People at Risk of Cardiovascular Disease (TLC)
Brief Title: Tools for Lasting Lifestyle Changes
Acronym: TLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1100
Record Dates: First submitted 2018-11-16; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Diseases; Lifestyle Risk Reduction
Keywords: Primary intervention
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 'Lifestyle counselling and exercise' . (Experimental): The study is a single-arm study where all participants undergo the same intervention 'Lifestyle counselling and exercise' .
  Interventions: Behavioral: Lifestyle counselling and exercise

INTERVENTIONS:
Behavioral: Lifestyle counselling and exercise — The program consists of:
  1. Instructor-led training twice a week,
  2. One individual nutritionist counselling session of followed by three group based two-hour nutritionist counselling focusing on practical food purchase and preparation and
  3. Three two-hour psychologist-led group counselling sessions based on implementation intentions theory and practical help to make if-then plans focusing on changing food and activity habits.

SUMMARY:
Pilot and feasibility study; a complex intervention focusing on lifestyle change to increase physical activity and reduce cardiovascular disease (CVD) risk among high risk individuals.

DETAILED DESCRIPTION:
Interdisciplinary, mixed-method, prospective and single-arm exploratory study aimed to explore study feasibility, responsiveness, participants adherence and adverse events among the participants before deciding to proceed to full-scale evaluation.

Enrollment of max. 20 obese people (BMI>30) with sedentary lifestyle and increased CVD-risk (NORRISK2)..

Participants general health status including cardiopulmonary fitness will be assessed both before and after the intervention (blood pressure, ECG, spirometry, treadmill tests VO2max, blood tests, body composition by Dual-energy X-ray absorptiometry (DEXA) measurements) Participants´ functional capacity assessed by several range of motion tests. Participants nutritional and psychological status assessed by validated questionnaires.

Several blood-tests and ECG will be recorded at three months.

Daily activity level during and six months after the intervention period monitored by Polar M430 pulse watch.

The participants will be interviewed with focus on their prior health, activity habits and intervention experiences at three months and six months after end of the intervention. Two focus-group interviews at end of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-74 years
2. BMI> 30
3. Moderate elevated NORRISK 2 score
4. Motivation for lifestyle change
5. Has agreed to attend and participate in a student study during the study period

Exclusion criteria: 1.External disease with short life expectancy 2.Diseases that limit physical activity in the project 3.Serious mental illness 4. Previous myocardial infarction 5.EKG changes that show severe rhythm disturbance, unstable angina or heart attack

5.EKG changes that show severe rhythm disturbance, unstable angina or heart attack:

Ages: 55 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline physical activity at 6 months | 6 months
  Change from baseline steps counted by activity trackers (Polar M430) at 6 months

SECONDARY OUTCOMES:
Change from baseline central obesity at 6 months | 6 months
  Change from baseline waist circumference (cm) at 6 months standardized measured
Change from baseline VO2max at 6 months | 6 months
  Change from baseline VO2max at 6 months measured on treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Sameline Grimsgaard, MD, MPH, PhD, Principal Investigator — Professor
Locations (1):
- UiT the Arctic University of Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deraas TS, Hopstock L, Henriksen A, Morseth B, Sand AS, Njolstad I, Pedersen S, Sagelv E, Johansson J, Grimsgaard S. Complex lifestyle intervention among inactive older adults with elevated cardiovascular disease risk and obesity: a mixed-method, single-arm feasibility study for RESTART-a randomized controlled trial. Pilot Feasibility Stud. 2021 Oct 27;7(1):190. doi: 10.1186/s40814-021-00921-0. PMID 34706777
- [Derived] Hopstock LA, Deraas TS, Henriksen A, Martiny-Huenger T, Grimsgaard S. Changes in adiposity, physical activity, cardiometabolic risk factors, diet, physical capacity and well-being in inactive women and men aged 57-74 years with obesity and cardiovascular risk - A 6-month complex lifestyle intervention with 6-month follow-up. PLoS One. 2021 Aug 25;16(8):e0256631. doi: 10.1371/journal.pone.0256631. eCollection 2021. PMID 34432850
- [Derived] Henriksen A, Sand AS, Deraas T, Grimsgaard S, Hartvigsen G, Hopstock L. Succeeding with prolonged usage of consumer-based activity trackers in clinical studies: a mixed methods approach. BMC Public Health. 2020 Aug 27;20(1):1300. doi: 10.1186/s12889-020-09406-w. PMID 32854671